CLINICAL TRIAL: NCT01331187
Title: Influence on Diagnostics and Inpatient Workflow of Routinely Adding Ultrasound Screening by Pocket-size Ultrasound in a Medical Department
Brief Title: Influence of Routinely Adding Ultrasound Screening in Medical Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Nord-Trøndelag HF (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LH-2011-1
Record Dates: First submitted 2011-03-30; First posted 2011-04-07 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Heart Disease; Dyspnea; Aortic Disease; Kidney Disease; Liver Disease
Keywords: Echocardiography; Heart failure; Ultrasonography; pocket-size device; Aorta; Education
MeSH Terms: conditions — Heart Diseases; Dyspnea; Aortic Diseases; Kidney Diseases; Liver Diseases; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (Active Comparator): Usual care diagnostics. No routinely ultrasound examination
  Interventions: Other: Usual care
- Routinely ulasonography (Experimental): Patients will routinely be examined with ultrasound at admittance in addition to usual care diagnostics
  Interventions: Procedure: Pocket-size ultrasonography

INTERVENTIONS:
Procedure: Pocket-size ultrasonography — Routinely adding a ultrasound examination of the heart, pleura, great abdominal vessels, liver/gall bladder and kidneys at patients admittance to hospital
  Arms: Routinely ulasonography
Other: Usual care — No intervention, except for usual care (goal-directed diagnostics)
  Arms: Usual care

SUMMARY:
Ultrasound (US) is widely used as a diagnostic tool in a hospital setting. In a medical department, diagnosis like heart failure or most kinds of heart diseases, hypervolemia, hypovolemia, pleural effusion, pericardial effusion, ascites, diseases in the gall bladder/bile tract, urine tract and venous thrombosis are common. US is the key diagnostic tool in these diagnosis, and on early diagnosis is crucial with respect to the patients well-being and inpatients workflow.

1. The aim is to study the clinical use of pocket-size US as a screening diagnostic tool in an medical department with respect to inpatients workflow and diagnostics.

Method: Patients admitted (in certain preset periods) to Department of medicine will be randomized to routinely adding an ultrasound examination with pocket-size device by residents on call. Time to definitive diagnosis, time to definitive treatment and time to discard will be recorded. US findings will be validated against standard echocardiography, or standard US/CT/MRI performed at the Radiological department.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Dep. of Medicine at Levanger Hospital

Exclusion Criteria:

* Not able to give informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Time to definitive diagnosis | 3 months
  Time from admittance to definitive diagnosis

SECONDARY OUTCOMES:
Test-retest reproducibility | 3 months
  Pocket-sized ultrasound recordings by residents will be validated against reference methods (echocardiography and radiologic examinations by sepcialists)to assess sensitivity, specificity, positive and negative predictive values of pocket-size ultrasound.
Diagnostic outcome of additional ultrasound examination according to educational level of the performer | 3 months
  Study the diagnostic outcome of ultrasound screening related to the educational level and skills of the user
Time to definitive treatment | 3 months
  Time from admittance to definitive treatment
Time to discharge | 3 months
  Time from patients admittance to discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: Havard Dalen, MD, PhD, Study Chair — Levanger Hospital/Norwegian University of Science an Technology
Locations (1):
- Department of Medicine, Levanger Hospital, Nord-Trøndelag Health Trust, Levanger, Norway

REFERENCES:
- [Background] Sicari R, Galderisi M, Voigt JU, Habib G, Zamorano JL, Lancellotti P, Badano LP. The use of pocket-size imaging devices: a position statement of the European Association of Echocardiography. Eur J Echocardiogr. 2011 Feb;12(2):85-7. doi: 10.1093/ejechocard/jeq184. Epub 2011 Jan 7. PMID 21216764
- [Background] Prinz C, Voigt JU. Diagnostic accuracy of a hand-held ultrasound scanner in routine patients referred for echocardiography. J Am Soc Echocardiogr. 2011 Feb;24(2):111-6. doi: 10.1016/j.echo.2010.10.017. Epub 2010 Dec 3. PMID 21126857
- [Background] Roelandt JR. Ultrasound stethoscopy. Eur J Intern Med. 2004 Oct;15(6):337-347. doi: 10.1016/j.ejim.2004.08.002. PMID 15522567
- [Background] Kimura BJ, Shaw DJ, Agan DL, Amundson SA, Ping AC, DeMaria AN. Value of a cardiovascular limited ultrasound examination using a hand-carried ultrasound device on clinical management in an outpatient medical clinic. Am J Cardiol. 2007 Jul 15;100(2):321-5. doi: 10.1016/j.amjcard.2007.02.104. Epub 2007 May 29. PMID 17631091
- [Background] Lucas BP, Candotti C, Margeta B, Evans AT, Mba B, Baru J, Asbury JK, Asmar A, Kumapley R, Patel M, Borkowsky S, Fung S, Charles-Damte M. Diagnostic accuracy of hospitalist-performed hand-carried ultrasound echocardiography after a brief training program. J Hosp Med. 2009 Jul;4(6):340-9. doi: 10.1002/jhm.438. PMID 19670355
- [Background] Martin LD, Howell EE, Ziegelstein RC, Martire C, Whiting-O'Keefe QE, Shapiro EP, Hellmann DB. Hand-carried ultrasound performed by hospitalists: does it improve the cardiac physical examination? Am J Med. 2009 Jan;122(1):35-41. doi: 10.1016/j.amjmed.2008.07.022. PMID 19114170
- [Background] Moore CL, Copel JA. Point-of-care ultrasonography. N Engl J Med. 2011 Feb 24;364(8):749-57. doi: 10.1056/NEJMra0909487. No abstract available. PMID 21345104